CLINICAL TRIAL: NCT01912690
Title: The Influence of Different Training Regimens on Electrical Stability Following Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TRAINING
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-08

CONDITIONS: Ischemic Heart Disease; Congestive Heart Failure
MeSH Terms: conditions — Myocardial Ischemia; Heart Failure | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- standard of care (Placebo Comparator)
- aerobic training only (Active Comparator)
  Interventions: Other: aerobic training
- Aerobic and strength training (Active Comparator)
  Interventions: Other: aerobic and strength training

INTERVENTIONS:
Other: aerobic training
  Arms: aerobic training only
Other: aerobic and strength training
  Arms: Aerobic and strength training

SUMMARY:
The hypothesis of the study is that aerobic conditioning following acute heart attack will improve autonomic function and electrical stability of the heart.

ELIGIBILITY:
Inclusion Criteria:

* s/p acute myocardial infarction 14-30 days
* ability to perform exercise

Exclusion Criteria:

* unstable angina
* chronic atrial fibrillation
* severely reduced LV function
* NYHA 4
* severe valvular disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Left ventrcular dyssynchrony | 3 months
  Assessed by 2-D strain imaging

SECONDARY OUTCOMES:
Autonomic function | 3 months
  Assessed by Holter

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah University Medical Center, Jerusalem, Israel